CLINICAL TRIAL: NCT07094789
Title: Assessment of Safety and Feasibility of Focused Ultrasound Next Generation Dome Helmet (NGDH) to Perform Neuromodulation in Patients With Treatment-Resistant Depression
Brief Title: Focused Ultrasound Neuromodulation in Patients With Treatment-Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6702
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Treatment-Resistant Depression; Treatment-resistant Depression (TRD)
Keywords: Neuromodulation; Focused Ultrasound; Treatment-Resistant Depression; FUS; TRD; CSTC Circuit
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focused Ultrasound Neuromodulation (Experimental): Participants will receive two sessions of Magnetic Resonance-guided focused ultrasound neuromodulation targeting regions within the cortical-striatal-thalamic circuit (CSTC) implicated in treatment-resistant depression. Treatments will be spaced four weeks apart. All participants will receive the same intervention and will be followed for 4 weeks post-treatment to evaluate clinical outcomes, adverse events, and depression symptoms.
  Interventions: Device: Next Generation Dome Helmet (NGDH)

INTERVENTIONS:
Device: Next Generation Dome Helmet (NGDH) — Participants will receive two sessions of Magnetic Resonance-guided focused ultrasound neuromodulation, spaced four weeks apart, using the Next Generation Dome Helmet device. Treatments will target regions within the CSTC circuit identified by advanced MRI scans. Each session will include pre-treatment assessments, precise sonications of deep brain structures, real-time safety monitoring, and post-treatment imaging.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and initial effectiveness of Magnetic Resonance-guided focused ultrasound neuromodulation using the Next Generation Dome Helmet (NGDH) device in patients with treatment-resistant depression. This is a prospective, single-arm, non-randomized study.

Participants will:

* Undergo two focused ultrasound treatment sessions targeting nodes of the cortical-striatal-thalamic circuit (CSTC) , spaced four weeks apart.
* Return for follow-up visits at 24 hours, 2 weeks, and 4 weeks after each treatment session, during which clinical scales and imaging assessments will be conducted to monitor safety and clinical effects.

DETAILED DESCRIPTION:
A total of 20 participants with treatment-resistant depression will be enrolled and treated in this study. Participants will be recruited through local psychiatric practices, referrals from participating institutions, and external referrals, including both physician and self-referrals.

Eligibility will be assessed during a dedicated screening appointment conducted by the study coordinator in collaboration with a study-affiliated physician. The anticipated enrollment period is approximately two years, beginning from the date of first patient enrollment to the enrollment of the final participant.

ELIGIBILITY:
Inclusion Criteria:

1. Deemed to have the capacity to provide informed consent.
2. Aged between 18 and 65 years.
3. Diagnosis of major depressive disorder (MDD) according to DSM-5 criteria.
4. Total score >20 on the Hamilton Depression Rating Scale (HAMD-17).
5. On a stable regimen of psychiatric medications for at least 30 days prior to enrollment.
6. Documented previous trial of at least two first-line antidepressant agents at adequate dose and duration, as assessed by two psychiatrists.
7. Documented previous trial of cognitive behavioral therapy (CBT) or psychotherapy for MDD, sustained for at least 6 weeks.

Exclusion Criteria:

1. Pregnant or intending to become pregnant during the study period.
2. Diagnosis of a substance use disorder (excluding cannabis or nicotine) of moderate severity or greater, or when the substance is the primary focus of treatment, based on DSM-5 criteria.
3. Known active seizure disorder, significant head injury with an imaging-verified lesion
4. Unstable medical illness.
5. Not eligible for 3-Tesla MRI (i.e. MRI-incompatible pacemaker)
6. Inability to reliably attend required screening, treatment, or follow-up appointments.
7. Severe claustrophobia, as identified by the participant, that would prevent completion of MRI procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety and Feasibility of FUS Next Generation Dome Helmet (NGDH) to Perform Neuromodulation in Patients with Treatment-Resistant Depression | Assessments will be conducted at the baseline visit, 24 hours after the first treatment, 2 weeks after the first treatment, 24 hours after the second treatment, and at 2 and 4 weeks following the second treatment.
  Assessment of the frequency and severity of adverse events associated with focused ultrasound neuromodulation in patients with treatment-resistant depression using the Next Generation Dome Helmet device. Adverse events, including procedure-related complications and neurological events, will be documented and assessed throughout the study period.

SECONDARY OUTCOMES:
Clinical Efficacy - Change in Depressive Symptoms measured by Hamilton Depression Rating Scale (HAMD-17) | Assessed at 2 weeks after first treatment and 2 and 4 weeks after second treatment.
  Clinical efficacy will be evaluated by analyzing changes in symptom scores using repeated-measures analysis of variance. The primary measure of clinical efficacy will be the Hamilton Depression Rating Scale (HAMD-17) score.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No